CLINICAL TRIAL: NCT04763499
Title: The Influence of Daily Strawberry Intake on Vascular Health in Elderly Men
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruiting progress
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1567320
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Vascular Dilation
Keywords: strawberry, diet, vascular function, inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, crossover dietary intervention trial.
Who Masked: Participant, Investigator
Masking Description: both the control and freeze dried strawberry powders are package with only a code as the identifier
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze dried strawberry powder (Experimental): 39g of freeze dried strawberry powder, which represents three daily servings of strawberries.
  The powder will be mixed in one cup of water.
  Interventions: Other: freeze dried strawberry powder
- control powder (Placebo Comparator): 39 g of a powder that matches the sugar and caloric content of the experimental powder. The powder will be mixed in one cup of water.
  Interventions: Other: freeze dried strawberry powder

INTERVENTIONS:
Other: freeze dried strawberry powder — approximately 24 strawberries that have been freeze dried into a powder

SUMMARY:
The overall objective of this proposed trial is to examine the vascular protective effects provided by the daily consumption of 39g of freeze dried strawberry powder (FDSP) for four weeks. The study population will be older men (60-80 years of age).

DETAILED DESCRIPTION:
The proposed project will determine the influence of short-term FDSP intake on microvascular function in older men (60-80 years of age). The Framingham reactive hyperemia index (fRHI) will be used as a measure of microvascular function, and will be measured using peripheral arterial tonometry (PAT; EndoPAT200). Secondary outcomes will assess circulating levels of nitrate and nitrite, insulin-like growth factor (IGF), inflammatory cytokines, NADPH oxidase, platelet aggregation, plasma lipids and blood pressure. This suite of markers will provide insight on physiological outcomes and risk factors associated with CVD development, and the metabolic and signaling pathways that influence them. To accomplish the above, after a 4 week run in period of no powder intake, twenty men (60-80 years of age) will be randomly assigned to consume 39 g of FDSP or a control powder for four weeks in a randomized, double-blind, controlled crossover study. This study design will compare the short-term (four week) response of FDSP intake to an isocaloric control powder that provides no polyphenols, as well as to their habitual diet where no powder was consumed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 25.0 - 35 kg/m2

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Visit 1 Reactive Hyperemia Index (RHI; EndoPAT 2000) ≥ 2.8
* Dislike or allergy strawberries
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Prescription medications other than on a 6 month self-reported stable dose of medications for lipid lowering and/or hypertension.
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Fruit consumption ≥ 3 cups/day
* Regular consumption of strawberries (2-3 servings/week)
* Vegetable consumption ≥ 4 cups/day
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Peripheral artery disease Raynaud's syndrome or disease
* Inability to properly place or wear the PAT probes or abnormal measurements on pre- screening PAT
* Abnormal Metabolic or CBC panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Supplement use other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Cannabis use
* Current enrollee in a clinical research study.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Framingham Reactive Hyperemia Index (fRHI) | 4 weeks
  fRHI as a measure of microvascular function will be measured by peripheral arterial tonometry (PAT).

SECONDARY OUTCOMES:
platelet aggregation | 4 weeks
  optimal platelet aggregometry using collagen and adp as agonist
Th17 cytokines | 4 weeks
  TH17 Luminex panel: Interleukin (IL)-1b, IL-4, IL-6, IL-10, IL-17a, IL-21, IL-22, IL-23, IL-31, IL-33, IFNgamma, TNFalpha, IL-17f.
insulin like growth factor (IGF) and binding proteins (IGFBP) | 4 weeks
  Luminex panel: IGF-1, -2 and IGFBP 1-7
Nicotinamide adenine dinucleotide phosphate (NADPH) oxidase | 4 weeks
  soluble form marker of oxidative stress
total nitrate and nitrite | 4 weeks
  plasma total nitrate and nitrite

OTHER OUTCOMES:
blood pressure | 4 weeks
  systolic and diastolic blood pressure
plasma lipids | 4 weeks
  clinical lipid panel

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — Professor of Nutrition and Internal Medicine
Locations (1):
- University of California, Davis; Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/are-you-a-man-between-60-and-80-years-old-help-us-learn-about-how-strawberries-influence-your-health-423731/